CLINICAL TRIAL: NCT04333290
Title: Phase 1 Study Evaluating the Safety of [11C]MeDAS Myelin-Targeting PET Agent in Humans
Brief Title: Study Evaluating the Safety of Myeliviz Myelin-Targeting PET Agent
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unable to obtain Myeliviz for trial
Sponsor: Robert Fox (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Sponsor-Investigator, Robert Fox, Vice Chair, Research, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MeDAS-001
Record Dates: First submitted 2020-03-18; First posted 2020-04-03 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: myelin; PET; central nervous system; brain; spinal cord; demyelination; MRI
MeSH Terms: conditions — Demyelinating Diseases | interventions — N-methyl-4,4'-diaminostilbene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm: Healthy subjects (Experimental): The PET radiotracer Myeliviz ([11C]MeDAS) will be administered to healthy subjects twice and PET scans will be obtained each time. This will allow assessment of the PET image quality, PET scan reproducibility and radiotracer distribution.
  Interventions: Drug: [11C]MeDAS

INTERVENTIONS:
Drug: [11C]MeDAS — PET radiotracer
  Other Names: Myeliviz

SUMMARY:
This study evaluates the safety of [11C]MeDAS, a PET radiotracer.

DETAILED DESCRIPTION:
Myelin PET imaging provides a new type of information regarding the integrity of the central nervous system based on molecular imaging of myelin. Preclinical studies have shown [11C] MeDAS uptake in the brain and spinal cord to be an indicator of the microstructural integrity of the tissue.

[11C]MeDAS PET (Positron Emission Tomography) scans will be performed on healthy subjects at 2 timepoints to assess for safety of the radiotracer and to assess its performance in humans. Following measurement of [11C]MeDAS pharmacokinetics and biodistribution, an optimal protocol for dosing and imaging will be established.

ELIGIBILITY:
Inclusion Criteria:

* Subject reports no known physical diseases of the central nervous system including no history of mental health disorders.
* Capable of giving informed consent
* Efforts will be made to include approximately equal numbers of women and men. Efforts will be made to include individuals of diverse ethnicities, as reflected in the local clinic population.

Exclusion Criteria:

* Age <18 or >65
* History of malignant hypertension or hypertensive crisis
* Known infectious disease requiring treatment during the course of the study
* Subject reported history of substance abuse
* inability to undergo an MRI or PET scan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Radiation dosimetry | Less than or equal to 2 hours
  Whole body radiotracer uptake, as measured using PET scan image data. Radiotracer uptake will be measured in absolute counts and using distribution volume ratios.
Biodistribution analysis | Less than or equal to 2 hours
  Organ-specific radiotracer uptake, as measured using PET scan image data. Radiotracer uptake will be measured in absolute counts and using distribution volume ratios.
Metabolism analysis | Less than or equal to 2 hours
  Analysis of in vivo radiotracer metabolism using liquid chromatography, with quantification of relative peak areas under the curve.
Pharmacokinetic analysis based on PET scan data | Less than or equal to 2 hours
  Determination of time-dependent radiotracer distribution using PET scan image data, with time measurement in minutes, PET data measured in absolute counts, and position in the body determined by organ segmentation.
Analysis of time-dependent radiotracer distribution based on arterial blood sampling | Less than or equal to 2 hours
  Determination of time-dependent radiotracer distribution as assessed by arterial blood sampling, using scintillation counting for determination of radiotracer activity. Time is measured in minutes and radiotracer quantity is assayed by scintillation counting with units in absolute counts.

SECONDARY OUTCOMES:
Brain imaging characterization | Less than or equal to 2 hours
  Analyze patterns of radiotracer distribution in the brain using PET scan image data. This is an intrinsically qualitative analysis and image data will be assessed by visual inspection. Based on findings of this first-in-human study, preliminary quantitative assessment using coregistration with structural imaging, anatomic segmentation and partial volume correction will be performed to calculate distribution volume ratios for areas of interest.
Spinal cord imaging characterization | Less than or equal to 2 hours
  Analyze patterns of radiotracer distribution in the spinal cord using PET scan image data. This is an intrinsically qualitative analysis and image data will be assessed by visual inspection. Based on findings of this first-in-human study, preliminary quantitative assessment using coregistration with structural imaging, anatomic segmentation and partial volume correction will be performed to calculate distribution volume ratios for areas of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Fox, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
data will be available per NIH policies